CLINICAL TRIAL: NCT03017638
Title: Analgesic Efficacy of Quadaratus Lumborum Block (QLB) for Laparoscopic Colectomy Surgery: A Prospective Observational Case Control Trial to Evaluate Clinical Outcomes
Brief Title: Analgesic Efficacy of Quadaratus Lumborum Block (QLB) for Laparoscopic Colectomy Surgery: A Prospective Case Control Trial to Evaluate Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0832-16
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2017-01

CONDITIONS: Block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients receiving QLB and questionaires: Patients undergoing primary laparoscopic colectomy patients under general anesthesia with an additional Quadratus lumborum block (QLB ) will be asked to fill out a questionnaires detailing: numeric verbal analogue scores (VAS) and quality of recovery score(QoR) preoperatively, 24 hours and 48 hours and four weeks after surgery. Additional data will be collected: ASA physical status, demographics, intra- and post operative opiate(expressed as morphine equivalent in mg/kg) and non opiate consumption in order to assess the analgesic efficacy of QLB for primary laparoscopic colectomy. QLB will be performed as per standard routine regimens, in the operating room after induction of general anesthesia and prior to surgery.
  Interventions: Other: Questionaire
- Historical control: The control subjects' data will be assessed reviewing patient records. Data will include:
  * Maximal PACU VAS pain score (per nursing charts)
  * Overall POD 24 hours and 48 hours and 4 weeks opioid consumption (overall morphine mg/kg equivalent dose)
  * POD 24 and 48 hours and 4 weeks Respiratory complications

INTERVENTIONS:
Other: Questionaire — Patients undergoing primary laparoscopic colectomy patients under general anesthesia with an additional Quadratus lumborum block (QLB ) will be asked to fill out a questionnaires detailing: numeric verbal analogue scores (VAS) and quality of recovery score(QoR) preoperatively, 24 hours, 48 hour and four weeks after surgery. Additional data will be collected: ASA physical status, demographics, intra- and post operative opiate(expressed as morphine equivalent in mg/kg) and non opiate consumption in order to assess the analgesic efficacy of QLB for primary laparoscopic colectomy. QLB will be performed as per standard routine regimens, in the operating room after induction of general anesthesia and prior to surgery.
  Groups: Patients receiving QLB and questionaires

SUMMARY:
Pain after abdominal surgery can be extensive. Pain control is an important component of patient comfort and participation in rehabilitation. Multimodal analgesia methods have shown to reduce postoperative pain, and have been addressed to be a crucial part of the Enhanced Recovery after Surgery (ERAS) protocols.

Quadratus lumborum block (QLB) is a posterior abdominal wall block which analgesic efficacy has been shown for abdominal surgeries, and also for different laparoscopic procedures, such as ovarian surgery.

The aim of this study is to assess QLB's analgesic efficacy for laparoscopic colectomy surgeries, using serial pain score assessments and overall opioid consumption; its effect on patient satisfaction; and its effect on the development of postoperative respiratory complications. This study is a prospective clinical trial assessing the effect of application of QLB as a regional analgesic technique for primary laparoscopic colectomy, in comparison to a historical retrospective cohort.

DETAILED DESCRIPTION:
A. Specific Aims Pain control is an important component of patient comfort and rehabilitation after surgery. The aim of the study is to improve multimodal analgesia and reduce postoperative pain for laparoscopic colonic surgery. We hypothesize that performing a Quadratus Lumborum Block (QLB) prior to start of laparoscopic colon surgery will provide significant analgesic effect. As such, the primary endpoint of this study is the patient's maximal reported pain scores using a numeric verbal analogue scale (1-10) elicited during the patient's post operative recovery unit (PACU) stay, 24 hours, 48 hours and 4 weeks after surgery.

Secondary endpoints are:

* Total opioid consumption during PACU stay and on 24 hours ,48 hours and 4 weeks after surgery.
* Length of hospital stay
* Overall patient satisfaction - will be documented on 24 hours after surgery, 48 hours and 4 weeks after surgery.
* Minimal saturation during PACU stay
* Development of postoperative respiratory complications until patient discharge: re-intubation, documented apneas, severe hypoxemia (measured saturations <94%; or arterial blood oxygen partial pressure in relation to inspired oxygen concentration [PaO2/FiO2] ration below 200)

Research Design and Methods The study is a prospective clinical trial assessing the effect of application of QLB as a regional analgesic technique for primary laparoscopic colectomy, in comparison to a historical cohort.

Inclusion Criteria:

All primary laparoscopic colectomy patients are eligible for inclusion in the study.

Exclusion criteria are:

* Allergy to local anesthetics or to systemic opioids
* Contraindication to regional anesthesia technique, such as local infection or coagulopathy
* Requirements of more than 30 mg morphine equivalent daily prior to surgery
* ASA IV or greater
* Psychiatric or cognitive disorders
* Incarceration
* Renal insufficiency with Cr > 2.0
* Hepatic failure
* Pregnancy
* Age under 18 years Potential risks for the procedure, which will be explained to the patient, include: bleeding, local infection, local anesthetic toxicity. All are commonly listed as rare complications of the procedures.

After consenting to participation, QLB will be placed in the operating room after induction of general anesthesia and prior to surgery.

For participating patients, the following data will be collected by the research staff: ASA physical status, age, height, weight, gender, intra- and post operative quantitative opiate use (expressed as morphine equivalent in mg/kg), numeric VAS scores, and QoR score (form included).

Intraoperative care:

Intraoperative anesthesia will be achieved using a general anesthetic technique. Intraoperative analgesia will be administered per anesthesiologists' discretion.

All patients will have a laparoscopic colectomy. QLB Procedure Details Patients will lie in the supine position. Aseptic precautions will be taken by wearing a surgical cap, a mask, sterile gown and sterile gloves after disinfection of the hands. The abdominal region will be disinfected using chlorhexidine solution, and then covered in sterile drapes. A high frequency linear ultrasound (US) transducer (Philips 4-12L linear transducer with a frequency of 6-12 MHz, Milwaukee, WI) covered with sterile plastic sheath will be placed in the anterior axillary line to visualize the typical triple abdominal layers. Then, the probe will be withdrawn to the posterior axillary line, where at this juncture the layers of abdominal layers start to taper: the transversus abdominis muscle converging with the internal oblique and external oblique forming a singular aponeurosis, blending with the quadratus lumborum muscle, which inserts from the dorsal aspect of the body [Figure 1].

At the junction of the tapered ends of abdominal muscles and QL, and under continuous US guidance, a 22 gauge 80 mm insulated Tuohy needle (SonoPlexStimu, PAJUNK MEDIZINTECHNOLOGIE GEISINGEN, GERMANY) will be inserted in plane [Figure 2]. Its proper location will be verified using 0.9% NaCl injection. After position verification and following negative aspiration, 25 mL of 0.5% ropivacaine (Naropin-AstraZeneca, Sydney, North South Wales, Australia) will be injected under US visualization, in 3-5 mL aliquots, separated by repeated negative aspirations, meant to confirm absence of intravascular injection.

Post-operative analgesia All patients will be given a standard regimen of IV acetaminophen 1000mg q8hr, and IV Tramadone 100 mg q8hr (concurrent with prophylactic anti-emetic therapy using IV metoclopramide 10 mg q8hr), both started intraoperatively prior to conclusion of surgery, and continuing for 48 hours.

While in PACU, all patients will be administered a morphine patient controlled analgesia (PCA) infusion pump (Graesby 3300®, Smith Medical International Ltd. Watford, UK; IVAC® PCAM®, Cardinal Health Inc., Rolle, Switzerland), for at least 48 hours. Per institutional protocol, PCA will be connected after bolus loading of IV 0.1 mg/kg morphine in the PACU.

Data Collection Patients will be enrolled for the study either during the pre-operative surgical appointment, or upon admission to the hospital. Upon enrollment, patients will have a Pain Management Questionnaire (attached) and VAS pain scores (0-10; 0 indicating no pain; 10 indicating most excruciating pain imaginable) recorded, and have their pre-operative analgesic medication documented.

To assess the effect of analgesia in PACU, maximal VAS pain scores, as reported by the patient to the PACU nursing staff, will be recorded. On 24 hours, 48 hoursafter surgery, the patient will indicate their level of pain using Pain Management Questionnaire (attached) and VAS pain scores. The patients will also complete their Pain Management Questionnaire and maximal VAS pain scores at 4 weeks after surgery (using a telephone survey).

Quality of recovery will be assessed using the Quality of Recovery (QoR) score 8-9, documented on 24 hours, 48 hours (personally) and also at 4 weeks after surgery (using a telephone survey).

In addition to the aforementioned scores, total analgesic medication will be documented: total opioid consumption (expressed in morphine equivalents doses, mg/kg) and during PACU stay and on 24 hours , and at 4 weeks after surgery.

Respiratory complications will be assessed by any of these events documented in the patient's chart during the postoperative period until patient discharge: re-intubation, documented apneas, severe hypoxemia (measured saturations <94%; or arterial blood oxygen partial pressure in relation to inspired oxygen concentration [PaO2/FiO2] ration below 200, if measured).

The control subjects' data will be assessed reviewing patient records. Their data will include:

* Maximal PACU VAS pain score (per nursing charts)
* Overall 24 hours , 48 hours and 4 weeks opioid consumption (overall morphine mg/kg equivalent dose)
* POD 24 and 48 hours and 4 weeks Respiratory complications

ELIGIBILITY:
Inclusion Criteria:

All primary laparoscopic colectomy patients are eligible for inclusion in the study.

Exclusion Criteria:

* Previous abdominal surgery
* Allergy to local anesthetics or to systemic opioids
* Contraindication to regional anesthesia technique, such as local infection or coagulopathy, or patients receiving anticoagulation therapy with smaller specifications than listed in professional guidelines.
* Contraindication to the Quadratus lumborum block such as defects or interferences in the abdominal wall obstructing anatomical structure visibility.
* Requirements of more than 30 mg morphine equivalent daily prior to surgery
* ASA IV or greater
* Psychiatric or cognitive disorders
* Incarceration
* Renal insufficiency with Cr > 2.0
* Hepatic failure
* Pregnancy
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults older than 18 years who are American Society of Anesthesiologists (ASA) Physical Status (PS) Classes 1-3. Inclusion criteria are patients undergoing primary laparoscop colectomy under general anesthesia with QLB.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-01-14 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Verbal analogue scale (VAS) | 24 Hours
  patient's maximal reported pain scores using a numeric verbal analogue scale (1-10) elicited during the patient's post operative recovery unit (PACU)
Verbal analogue scale (VAS) | 24 hours
  patient's maximal reported pain scores using a numeric verbal analogue scale (1-10) on postoperative day 1
Verbal analogue scale (VAS) | 48 hours
  patient's maximal reported pain scores using a numeric verbal analogue scale (1-10) on postoperative day 2

SECONDARY OUTCOMES:
Total opioid consumption in PACU | 24 hours
  Total opioid consumption during PACU stay
Total opioid consumption on postoperative day 1. | 24 hours
  Total opioid consumption on postoperative day 1.
Total opioid consumption postoperative day 2 | 48 hours
Total opioid consumption at four weeks postoperatively | 4 weeks
Length of hospital stay | 1 week
  Total days of hospitalization
Quality of recovery score (questionaire) four weeks postoperatively | 4 weeks
Quality of recovery score (questionaire) 1 day postoperatively | 24 hours
Quality of recovery score (questionaire) 48 postoperatively | 48 hours
Minimal saturation during PACU stay | 24 hours
Development of postoperative respiratory complications until patient discharge | 1 week
  re-intubation, documented apneas, severe hypoxemia (measured saturations <94%; or arterial blood oxygen partial pressure in relation to inspired oxygen concentration [PaO2/FiO2] ration below 200)

CONTACTS AND LOCATIONS:
Overall Officials: Shia Fein, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fischer HB, Simanski CJ, Sharp C, Bonnet F, Camu F, Neugebauer EA, Rawal N, Joshi GP, Schug SA, Kehlet H; PROSPECT Working Group. A procedure-specific systematic review and consensus recommendations for postoperative analgesia following total knee arthroplasty. Anaesthesia. 2008 Oct;63(10):1105-23. doi: 10.1111/j.1365-2044.2008.05565.x. Epub 2008 Jul 10. PMID 18627367
- [Result] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Result] O'Donnell BD, Iohom G. Regional anesthesia techniques for ambulatory orthopedic surgery. Curr Opin Anaesthesiol. 2008 Dec;21(6):723-8. doi: 10.1097/aco.0b013e328314b665. PMID 19009687
- [Result] Kang H, Ha YC, Kim JY, Woo YC, Lee JS, Jang EC. Effectiveness of multimodal pain management after bipolar hemiarthroplasty for hip fracture: a randomized, controlled study. J Bone Joint Surg Am. 2013 Feb 20;95(4):291-6. doi: 10.2106/JBJS.K.01708. PMID 23302898
- [Result] Kazak Bengisun Z, Aysu Salviz E, Darcin K, Suer H, Ates Y. Intraarticular levobupivacaine or bupivacaine administration decreases pain scores and provides a better recovery after total knee arthroplasty. J Anesth. 2010 Oct;24(5):694-9. doi: 10.1007/s00540-010-0970-x. Epub 2010 Jun 23. PMID 20571832
- [Result] Essving P, Axelsson K, Aberg E, Spannar H, Gupta A, Lundin A. Local infiltration analgesia versus intrathecal morphine for postoperative pain management after total knee arthroplasty: a randomized controlled trial. Anesth Analg. 2011 Oct;113(4):926-33. doi: 10.1213/ANE.0b013e3182288deb. Epub 2011 Aug 4. PMID 21821506
- [Result] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Result] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Result] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Result] Melvin JS, Stryker LS, Sierra RJ. Tranexamic Acid in Hip and Knee Arthroplasty. J Am Acad Orthop Surg. 2015 Dec;23(12):732-40. doi: 10.5435/JAAOS-D-14-00223. Epub 2015 Oct 22. PMID 26493971